CLINICAL TRIAL: NCT00837057
Title: A Randomized Controlled Multi-Center Trial of the Early Application of CRRT in Patients With Severe Sepsis or Septic Shock
Brief Title: Early Continuous Renal Replacement Therapies (CRRT) in Patients With Severe Sepsis or Septic Shock With Acute Kidney Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: sangbum hong, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: a085068
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-01

CONDITIONS: Severe Sepsis; Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Shock, Septic; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy; Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- early crrt, late crrt (Other)
  Interventions: Procedure: crrt

INTERVENTIONS:
Procedure: crrt — early CRRT (35 ml/kg/h)& acute kidney injury or failure or nearly anuria more than 2hr or late conventional dialysis indication
  Other Names: renal replacement therapy, timing

SUMMARY:
Severe sepsis or septic shock with acute kidney injury shows high mortality in intensive care unit. A few studies have shown CRRT relating the clinical improvement seems to be related to the early initiation of therapy. But there is no consensus for proper time of CRRT may improve the prognosis.

The study is a prospective randomized one center trial comparing two treatments in patients suffering from septic shock complicated with acute renal failure admitted to ICU, treated either early by CRRT (35 ml/kg/h) or by conventional RRT.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock (Bone criteria) for less than 14D
* RIFLE criteria : Injury or Failure or nearly anuria more than 2hr
* Age over 18 years
* Written informed consent by next of kin.

Exclusion Criteria:

* Cirrhosis child class C
* CRF or ESRD
* Too high APACHE II & SOFA score at admission
* Age over 80 years
* Life expectancy less than 3 months (metastatic cancer - hepatoma, lung ca.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Death from all causes at 28 days after randomisation | 28 day

SECONDARY OUTCOMES:
Death within the in the intensive care unit. Death within 90 days of randomisation. Death prior to hospital discharge. Length of ICU stay. The need for and duration of other organ support | 90 day

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787